CLINICAL TRIAL: NCT07143266
Title: Multidisciplinary Approach to Elucidate the Pathophysiology of Sleep Disorders in Patients With Hypothalamic and Pituitary Damage
Brief Title: Sleep Disorders in Hypothalamic and Pituitary Damage
Acronym: SDHPD
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-SUE-2024-36
Record Dates: First submitted 2025-06-17; First posted 2025-08-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Hypopituitarism; Sleep Wake Disorders; Hypothalamic Diseases; Oxytocin Deficiency
Keywords: Sleep Disorder; Oxytocin deficiency; Hypopituitarism; Hypothalamic damage
MeSH Terms: conditions — Hypopituitarism; Sleep Wake Disorders; Hypothalamic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hypopituitarism and hypothalamic damage with or without vasopressin deficiency: Differences between those patients with vasopressin deficiency (AVP-D) and those without AVP-D will be analyzed.
  Interventions: Other: This is an observational study. No drugs will be administered
- Healthy controls: Similar age, and BMI than the study group (patients with hypopituitarism) and matched by sex.
  Interventions: Other: This is an observational study. No drugs will be administered

INTERVENTIONS:
Other: This is an observational study. No drugs will be administered — Data from objective sleep evaluation (actigraphy, polisomnography and MLST), subjective sleep evaluation (questionnaires), neuroimaging (MRI and PET-CT), ophthalmological evaluation and hormone evaluation (urine and blood) will be collected in a cross-sectional manner, without performing any additional intervention.

SUMMARY:
Hypothalamus has a key role in multiple vital functions, including regulation of sleep-wake cycles. Oxytocin (OT), a neurohormone synthetized in the hypothalamus, has a wide range of physiological functions, including a putative role in improving sleep quality. Hypothalamic and pituitary damage (HPD) is associated with a clinically relevant OT deficient state and multiple and severe comorbidities including poor sleep quality, that have a well-known negative impact on general health and quality of life (QoL). Several factors may coexist in the pathophysiology of sleep disorders (SD) in HPD and SD might be a keystone in the persistence of some of the comorbidities observed in HPD. Therefore, appropriate identification and understanding of the mechanisms contributing to SD in HPD is mandatory to choose adequate preventive strategies and treatment. This project is aimed to (1) identify the prevalence of SD in HPD, (2) to determine OT role in sleep quality and (3) to identify potential mechanisms and mediators of sleep quality and their associations with clinical outcomes in patients with HPD with the ultimate goal of identifying preventive and therapeutic targets. We will use a controlled cross-sectional design of patients with HPD and sex-, BMI-, age- matched controls and an innovative cross-disciplinary approach bridging neuroendocrinology, psychology, neurophysiology, neuroimaging, nuclear medicine and neuroophthalmology disciplines to learn about the prevalence of SD in HPD and to disentangle the underpinning mechanisms behind SDs in HPD. The results of this project will be an extremely important step towards optimizing therapy for patients with HPD who have higher mortality and poor QoL despite appropriate hormone replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypothalamic-pituitary dysfunction (HPD) with at least one pituitary hormone deficiency and at least one clinical sign of hypothalamic damage (e.g., arginine-vasopressin deficiency (AVP-D) and/or severe obesity and/or hyperphagia; MRI suggestive of hypothalamic damage; traumatic brain injury; radiotherapy in the sellar region and/or brain tumors affecting the hypothalamus).
* Healthy controls matched for BMI, age, and sex.

Exclusion Criteria:

* Poor control of hormonal deficiencies in the previous 6 months.
* Use of new psychoactive drugs in the last 3 months or occasional use.
* Clinically significant liver, lung, kidney, and cardiovascular disease.
* Any neurological condition affecting brain function (stroke, dementia, uncontrolled epilepsy with recent seizures).
* Uncontrolled diabetes mellitus.
* Active psychosis.
* Ophthalmology: total blindness, Glaucoma, uveitis, visual acuity <0.6, or eye surgery in the previous 6 months.
* Any acute illness that the investigator determines may interfere with study participation or safety.
* Pregnancy or breastfeeding.
* Patients who refuse or are unable to provide written informed consent.
* In controls: presence of brain or pituitary tumor, radiation involving the hypothalamus or pituitary, and history of hypopituitarism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the Research Center for Pituitary Diseases and the Neurosurgery Department at the Hospital de la Santa Creu i Sant Pau, Barcelona, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disorders in patients with hypothalamic and pituitary damage compared to healthy controls | From enrollment to completion of the assessments at 3 months
  Prevalence (%) of patients with sleep disorders (assessed by objective and subjective measures of sleep):
  * Impaired sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI) and nocturnal polisomnography (PSG)
  * Daytime sleepiness assessed by Epworth Sleepiness Scale (ESS)
  * Obstructive Sleep Apnea (OSA) assessed by Berlin Questionnaire (BQ), Stop- BANG score risk and PSG
  * Insomnia assessed by Severity Index (ISI).
  * Daytime Sleepiness assessed by Multiple Sleep Latency Test (MSLT)

SECONDARY OUTCOMES:
Saliva oxytocin concentrations in patients compared to controls | From day 1 and day 2 of the objective sleep assessments (polisomnography and MSLT)
  * Oxytocin samples will be collected at 6:00 a.m., 12:00 p.m., 6:00 p.m., and 11:00 p.m.
  * Correlations between oxytocin concentrations and sleep disorders will be performed.
Urine 6-sulfametoxymelatonin concentrations in patients compared to controls | From day 1 and day 2 of the objective sleep assessments (polisomnography and MSLT)
  * Samples will be collected at 9:00 p.m., 6:00 a.m., 12:00 p.m., and 5:00 p.m in urine.
  * Correlations between 6-sulfametoxymelatonin concentrations and sleep disorders will be performed.
Prevalence of Brain structural and perfusion abnormalities using Magnetic Resonance Imaging in patients compared to controls | From enrollment to completion of the assessment at 3 months
  ROI related to sleep (e.g thalamus, cortex, amygdala) will be defined; gray matter hyperintensities will be quantified from the FLAIR image; DTI will calculate diffusor tensor parameters (FA, mean, axial and radial diffusivity) across the whole brain.
  Brain structural and perfusion abnormalities will be correlated with sleep measures
Prevalence of glucose brain metabolism abnormalities using Fluorodeoxyglucose Positron Emission Tomography in patients and controls | From enrollment to completion of the assessment at 3 months
  Glucose brain metabolism will be quantified at ROI. Brain glucose metabolism will be correlated with sleep measures
Prevalence of patients with neuroophthalmological damage (in patients with HPD only) assessed by an expert neuro-ophthalmologist | Baseline
  Prevalence (%) of patients with the following:
  * Impaired visual actuity
  * Impaired intraocular pressure using applanation tonometry
  * Impaired macular volume and retinal ganglion cell layer using standard Automated 24-2 Humphrey perimetry and spectral- domain optical coherence tomography (SD- OCT).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Aulinas, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain